CLINICAL TRIAL: NCT03246477
Title: Evaluation of the Long-term Impact of Maxillomandibular Advancement Osteotomy on Patients With Obstructive Sleep Apnea Syndrome
Brief Title: Long-term Impact of Maxillomandibular Advancement Osteotomy on Sleep Apnea Patients
Acronym: MIMOSA
Status: Completed | Type: Observational
Sponsor: AZ Sint-Jan AV (Other)
Collaborators: University Hospital, Ghent (Other)
Responsible Party: Principal Investigator, Nathalie Neyt, maxillofacial surgeon, principal investigator, AZ Sint-Jan AV
Other Study IDs: 2016/0876
Record Dates: First submitted 2017-02-10; First posted 2017-08-11 (Actual); Last update posted 2019-02-15 (Actual); Status verified 2019-02

CONDITIONS: Obstructive Sleep Apnea
Keywords: maxillomandibular advancement osteotomy; long-term results; quality of life; polysomnographic measurements; skeletal stability
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Background Maxillomandibular advancement surgery (MMA) has demonstrated high success rates, improving both the apnea-hypopnea index and associated patient' quality of life (QOL), in patients diagnosed with obstructive sleep apnea syndrome (OSAS). However, clinical relapse has been described in the target population, especially when associated with significant weight gain. Literature reporting the long-term impact of MMA for OSAS is lacking. The surgeons of the Division of Maxillofacial Surgery already started to perform this type of surgery in 1995.

Objectives The investigators aim to evaluate the long-term (minimum 15 years post-surgery) biologic and QOL impact of MMA in patients with OSAS. The biologic impact refers to the stability of hard and soft tissues and polysomnographic results.

Study design Retrospective study Both pre- en postoperative clinical imaging, polysomnography and quality of life questionnaires will be retrieved from all patients that were surgically treated with an MMA by one surgeon (CDC) between 01/11/1995 and 01/12/1999.

Conclusion Short-term data have shown high success rates for MMA in OSAS patients. However, long-term data are lacking. This retrospective study might provide us with more information about the incidence of clinical relapse fifteen to twenty years after surgery.

ELIGIBILITY:
Inclusion Criteria:

* clinically confirmed diagnosis of OSAS
* treated with an MMA between 01/11/1995 and 01/12/1999 by one surgeon (CDC)

Exclusion Criteria:

* not following abovementioned criteria

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients (n=10/12) with a clinically confirmed diagnosis of OSAS, that were treated with an MMA between 01/11/1995 and 01/12/1999 by one surgeon (CDC)
Sampling Method: Non-Probability Sample
Enrollment: 12 (Actual)
Dates: Start 2016-09 (Actual); Primary Completion 2017-12-31 (Actual); Study Completion 2017-12-31 (Actual)

PRIMARY OUTCOMES:
apnea-hypopnea index, as determined through polysomnography | minimum 15 years postoperative
oxygen saturation values, as determined through polysomnography | minimum 15 years postoperative

SECONDARY OUTCOMES:
evolution of patient quality of life, through Epworth Sleepiness Scale | preoperative
Stability of hard and soft head and neck tissue, according to manual anthropometry | min 15 years postoperative
Evolution of apnea-hypopnea index, as determined through polysomnography | preoperative
Evolution of apnea-hypopnea index, as determined through polysomnography | immediately postoperative
oxygen saturation values, as determined through polysomnography | preoperative
oxygen saturation values, as determined through polysomnography | immediately postoperative
evolution of patient quality of life, through Epworth Sleepiness Scale | immediately postoperative
evolution of patient quality of life, through Epworth Sleepiness Scale | minimum 15 years postoperative
evolution of patient quality of life, through OSAS questionnaire | preoperative
evolution of patient quality of life, through OSAS questionnaire | immediately postoperative
evolution of patient quality of life, through OSAS questionnaire | minimum 15 years postoperative
evaluation of hard and soft head and neck tissue, according to cone-beam CT imaging | minimum 15 years postoperative

CONTACTS AND LOCATIONS:
Overall Officials: Nathalie Neyt, Principal Investigator — AZ Sint-Lucas Brugge

IPD SHARING:
Plan to Share IPD: No